CLINICAL TRIAL: NCT05689073
Title: A Conversational AI System to Enhance Knowledge About Vaccines and Promote Vaccination: A Randomized Controlled Trial
Brief Title: A Conversational AI System to Enhance Knowledge About Vaccines and Promote Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2021KYPJ182
Record Dates: First submitted 2023-01-16; First posted 2023-01-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Vaccination Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversational AI system (Experimental)
  Interventions: Device: Conversational AI system
- Educational brochure (Active Comparator)
  Interventions: Other: Printed educational Brochure

INTERVENTIONS:
Device: Conversational AI system — The conversational AI system based on LLM processes user queries with a sophisticated generation, decision, action, and safety framework to provide optimal feedback. The system has several key features. Firstly, it utilizes retrieval-augmented in-context learning to enhance responses generated by the LLM, sourcing information from trustworthy websites. Secondly, it includes Guardrail module that addresses potential harmful content in the LLM-generated responses by clarifying and validating the content before delivery. Furthermore, the AI system is equipped with Self-checking memory module that retains essential clinical characteristics across multi-turn dialogues, ensuring the continuity and consistency of its interactions with users. The educational content about vaccination was derived from the official website of World Health Organization (https://www.who.int/news-room/questions-and-answers/item/vaccines-and-immunization-what-is-vaccination).
  Arms: Conversational AI system
Other: Printed educational Brochure — A printed brochure whose content about vaccination was derived from the official website of World Health Organization (https://www.who.int/news-room/questions-and-answers/item/vaccines-and-immunization-what-is-vaccination).
  Arms: Educational brochure

SUMMARY:
This study is designed to contribute to the growing body of evidence on the efficacy of digital health interventions. By rigorously evaluating the impact of the AI system on vaccine knowledge and acceptance, the study aims to inform future health communication strategies and policies. It stands as a potential model for integrating AI into public health initiatives, showcasing how technology can be harnessed to improve health outcomes on a large scale.

ELIGIBILITY:
Inclusion Criteria

* Individuals aged 18 or above
* Owning a smartphone/tablet capable of using the study app
* Willing to provide informed consent.

Exclusion Criteria

* Individuals with ocular or hearing disorders that preclude the use of mobile phones or reading.
* Individuals with mental disorders that preclude the use of mobile phones or reading.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptance of vaccines | Day 14
  Vaccine acceptance was evaluated based on responses to the question, 'Based on your actual situation, please choose the extent of your willingness to get vaccinated.' The response options were: Absolutely refuse, Refuse but uncertain about the future, Have not considered it yet, Accept but still considering, and Completely willing. Vaccine acceptance was considered if the participant selected 'Completely willing.

SECONDARY OUTCOMES:
Hesitancy of vaccination | Day 14
  The Vaccine Hesitancy Scale was developed based on the "3Cs" model (confidence, complacency, and convenience) by the SAGE Working Group on Vaccine Hesitancy, encompassing three aspects: confidence, complacency, and convenience. It utilizes a Likert 5-point scale (Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree) for scoring. For the complacency dimension, aspect, scoring is reversed with "Strongly Agree" to "Strongly Disagree" rated as 5 to 1 points, respectively. In contrast, other items follow the standard scoring, where "Strongly Agree" to "Strongly Disagree" are scored from 1 to 5 points. Confidence is measured by perceived vaccine safety and efficacy. Complacency is assessed through perceived necessity of the vaccine and the severity of the preventable diseases. Convenience is evaluated by the perceived ease of transportation and appointment scheduling.

OTHER OUTCOMES:
Feelings of coercion | Day 14
  To assess feelings of coercion related to vaccination, participants were asked a single question: 'When deciding whether to receive the vaccines, do you feel forced to either take or not take the vaccine?' This question utilizes a 5-point Likert scale (very low, low, neutral, high, very high) with lower scores indicating lower feelings of perceived coercion.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No